CLINICAL TRIAL: NCT06209593
Title: Acceptability (including Gastrointestinal Tolerance and Compliance) of a Plant Based High Energy Adult Enteral Formula
Brief Title: Acceptability and Tolerance Study of a Plant-based Tube Feed
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: PB 001
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Nutrition Disorders
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients well established on tube feeds will act as their own control: Each participant will receive the new trial feed a nutritionally complete standard enteral tube feed for a period of 7 days. The new trial feed is a food for special medical purposes for use under medical supervision. The Health Care Professional/ dietitian will determine the feeding regimen on an individual basis and the enteral formula will be provided via a feeding tube.
  Interventions: Dietary Supplement: Compleat plant protein tube feed

INTERVENTIONS:
Dietary Supplement: Compleat plant protein tube feed — Patients on a tube feed will act as their own control and switch to new tube feed.

SUMMARY:
This is a single arm, prospective, multi-centre study to evaluate the gastrointestinal tolerance and compliance over a 7-day period with a plant based tube feed.

DETAILED DESCRIPTION:
Enterally fed adults who are assessed by the Health Care Professional/dietitian as requiring an adult plant- based high-energy, enteral formula will be recruited. Data from 15 participants are required in order to submit an application to the UK Advisory Committee on Borderline Substances (ACBS) for product registration

ELIGIBILITY:
Inclusion Criteria:

* Patients 16 years and over and adults requiring a plant- based enteral tube feed (taking 50% or more of energy needs from their feeding tube) as part of their dietary management for disease related malnutrition
* Patients well-established and stable on current polymeric enteral tube feed.
* Willingly given, written, informed consent from patient

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator
* Under 16 years of age
* Patients on total parenteral nutrition
* Known food allergies to any ingredients including patients who have an allergy to milk protein e.g IgE and non- mediated as product contains traces of milk and allergy to peanuts due to the pea protein
* Patients with significant renal or hepatic impairment
* Participation in another interventional study within 2 weeks of this study.
* Patients with known or suspected ileus or mechanical bowel obstruction

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients established on a tube feed
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Baseline assessment and daily recording during intervention up to day 7 measuring Gastrointestinal tolerance | 7 days
  Diarrhoea, constipation, reflux, vomiting, wind, boating

CONTACTS AND LOCATIONS:
Overall Officials: James Evans, Principal Investigator — University College London Hospitals
Locations (1):
- Nu, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Will upload the data as it becomes available.